CLINICAL TRIAL: NCT06361134
Title: Efficacy of Supporting SAFE Early Intervention in the First Months of Life in Infants at Risk: A Randomized Controlled Trial
Brief Title: Efficacy of Supporting SAFE Early Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ayse Simsek, Gazi University, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14574941-302,08,01-
Record Dates: First submitted 2024-03-29; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2022-03

CONDITIONS: Infant Development; Physiotherapy; Early Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAFE Early Intervention Group (Experimental): A sensory-based, activity-focused early intervention program was implemented in an enriched environment (SAFE Early intervention). Children in the intervention group received home visits once a month and their families were coached. Families were informed about how to support their children. Home visits were made once a month for 10 weeks.
  Interventions: Behavioral: SAFE Early İntervention; Behavioral: NDT based therapy
- Control Group (Experimental): Home-based NDT program was applied to the control group. The babies in the group were examined in a clinic environment and the families were given booklets to support their children's development.
  Interventions: Behavioral: SAFE Early İntervention; Behavioral: NDT based therapy

INTERVENTIONS:
Behavioral: SAFE Early İntervention — As part of the intervention, sensory-based intervention was applied in an enriched environment. In the home setting, physiotherapists collaborated with the family to advance the intervention. The intervention was revised by making monthly home visits to infants with a corrected age of 42 weeks.
Behavioral: NDT based therapy — Neuromotor evaluations of the babies were performed in a clinical setting. The rehabilitation program to be implemented was given to the family as a booklet. The programs of the children examined in the clinic every month were revised.

SUMMARY:
Within the scope of the study, it was planned that risky babies would be treated with the SAFE early intervention approach for 10 weeks after they were discharged from the intensive care unit. Neurodevelopmental Treatment was applied to the control group. Sensory, motor and language development of the babies were evaluated before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

Neurologically and developmentally risky infant (such as premature birth, hypoxia, infection, hypoxic ischemic encephalopathy),

Having a NICU history of 15 days or more,

Exclusion Criteria:

congenital malformations, metabolic and genetic disease musculoskeletal system anomaly

Ages: 1 Month to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-05-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Test of Infant Motor Profile | 10 weeks
  High numerical scores indicate that infants notice and respond to stimuli less than their peers, meaning the infant is hypersensitive, while low numerical scores indicate that infants notice and respond to stimuli more than their peers, or are hypersensitive.

SECONDARY OUTCOMES:
Bayley Scales of Infant and Toddler Development, Third Edition, | 10 weeks
  Bayley Scales of Infant and Toddler Development- III is the most widely used tool for assessment of early development.Bayley-III including Cognitive, Language, and Motor scales . "1" if the child meets the scoring criteria for each item; If the child does not meet the criteria, he receives a score of "0". Raw scores for each subtest are summed (Total Raw Score) and then converted to scale scores, composite scores, percentile ranks and confidence intervals using the tables provided in the manual. These scores are used to determine the child's performance compared to norms from typically developing children their age (in months).
Infant/Toddler Sensory Profile 2 | 10 weeks
  The Infant/Toddler Sensory Profile (ITSP) was developed in response to the need for a standardized assessment of sensory processing for infants and toddlers. The ITSP is a caregiver questionnaire designed to measure in-fant/toddler responses to various sensory stimuli. It has two age bands: birth to6 (0-6) months and 7 to 36 (7-36) months, with 36 and 48 items, respectively. Each itemon the ITSP describes a certain behavior that may occur in daily life, with the fre-quency of such behaviors rated by the caregiver on a five-point Likert scale (1=always, 2=frequently, 3=occasionally, 4=seldom, and 5=never).
Infant/Toddler HOME Inventory | 10 weeks
  It is used to evaluate children's home environment. It evaluates the home environment of children aged 0-3 under six different subheadings. Parents rate the frequency of the child's behavior on a five-point scale from 1 (almost always) to 5 (almost never). The items in this test are; It evaluates six different areas: general, auditory, visual, tactile, vestibular and oral sensory processing. A higher score indicates that the answer occurs less frequently

CONTACTS AND LOCATIONS:
Locations (1):
- Erzurum Technical University, Erzurum, Turkey (Türkiye)

REFERENCES:
- [Derived] Yildiz A, Yildiz R, Apaydin U, Efkere PA, Gucuyener K, Hirfanoglu IM, Elbasan B. Effects of SAFE Early Intervention Approach in the First Months of Life in Infants at Risk: A Randomized Controlled Study. Child Care Health Dev. 2025 Jul;51(4):e70107. doi: 10.1111/cch.70107. PMID 40435392